CLINICAL TRIAL: NCT05250661
Title: Determination of the Effectiveness of Propolis in the Prevention of Oral Mucositis in Patients Receiving High Dose Chemotherapy: A Randomized Controlled Trial
Brief Title: Efficacy of Propolis in the Prevention of Oral Mucositis
Acronym: OM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Seher Çakmak, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E.6289
Record Dates: First submitted 2022-01-24; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; Propolis; High Dose Chemotherapy
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: Parallel group, two arm, prospective randomized controlled clinical trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqueous propolis extract (Experimental): The individuals in the intervention group were asked to gargle with 5 ml aqueous propolis extract four times a day after meals (morning, noon, evening and night before bedtime) and wait average one minute in the mouth and then spit, in addition to the standard practice of the clinic. According to the standard practice of the clinic, it was performed tanflex (3x1) and/or sodium bicarbonate (1x1) to the patients in the prevention of oral mucositis with the request of the physician. The patients were followed for 21 days. The 21-day period is consistent with the duration of mucositis healing in the literature. Follow-up and evaluation of patients who were discharged early were performed by home visits and made a phone call everyday.
  Interventions: Other: Aqueous propolis extract
- Control (No Intervention): Standard procedures of the clinic were applied to control group. According to the standard practice of the clinic, it was performed tanflex (3x1) and/or sodium bicarbonate (1x1) to the patients in the prevention of oral mucositis with the request of the physician. Follow-up and evaluation of patients who were discharged early were performed by home visits and made a phone call everyday.

INTERVENTIONS:
Other: Aqueous propolis extract — The patients gargled 4 times a day after meals and 5 ml each time. Patients were instructed to keep the propolis solution in their mouth for one minute, to touch all structures in the mouth, and not to eat or drink anything orally for one hour after spitting.
  Arms: Aqueous propolis extract

SUMMARY:
The study was carried out to determine the efficacy of propolis in the prevention of oral mucositis and gastrointestinal symptoms associated with oral mucositis in patients with leukemia, lymphoma, and myelodysplastic syndrome receiving high-dose chemotherapy and/or hematopoietic stem cell transplantation. 64 patients, 32 in the propolis and 32 in the control group, were involved in the prospective randomized controlled experimental study. While the standard oral care treatment protocol of the clinic was administered to the control group, aqueous propolis extract was applied to the propolis group in addition to the standard oral care treatment protocol.

DETAILED DESCRIPTION:
Objective: The study was carried out to determine the efficacy of propolis in the prevention of oral mucositis and gastrointestinal symptoms associated with oral mucositis in patients with leukemia, lymphoma, and myelodysplastic syndrome receiving high-dose chemotherapy and/or hematopoietic stem cell transplantation.

Study Design:

The study was conducted as a randomized controlled experimental study. Approval from the Ethics Committee and written permission from the Institution were obtained. After the participants were informed about the purpose of the study, their written consents were obtained. 64 patients, 32 in the propolis and 32 in the control group were involved in the study that was performed in the Hematology and Bone Marrow Transplantation Unit.

The control group patients used the standard oral care treatment protocol (Tanflex (3x1) and NaHCO3 (1x1)) of the clinic , while the propolis group used the aqueous extract of propolis in addition to this protocol. The individuals in the propolis group gargled 4 times a day (after meals and before going to bed at night) with 5 ml aqueous propolis extract. All patients underwent a daily intraoral examination up to 21 days from the start of high dose chemotherapy. Oral mucositis was recorded on the WHO oral toxicity scale and other gastrointestinal symptoms were recorded on the National Cancer Institute-Common Terminology Criteria for Adverse Events scale

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ability to communicate verbally
* Not having a diagnosed psychiatric disease
* Receiving inpatient high dose chemotherapy (diagnosed with leukemia, lymphoma and MDS)
* Hematopoietic Stem Cell Transplantation patients
* Zero OM score according to the World Health Organization Oral Toxicity Scale (WHOOTS)
* Karnofsky Performance Scale (KPS) score of 80 and above

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Time to onset of oral mucositis | For 21 days from the beginning of the chemotherapy
  Time to onset of oral mucositis was be evaluated by the World Health Organization Oral Toxicity Scale which record the extent and severity of oral mucositis every day.
  The World Health Organization Oral Toxicity Scale: range 0 to 4, Grade 0; none, Grade 1; mild, Grade 2; moderate, Grade 3; severe, Grade 4; life threatening
Incidence of oral mucositis | For 21 days from the beginning of the chemotherapy
  Incidence of oral mucositis was be evaluated by the World Health Organization Oral Toxicity Scale which record the extent and severity of oral mucositis every day.
  The World Health Organization Oral Toxicity Scale: range 0 to 4, Grade 0; none, Grade 1; mild, Grade 2; moderate, Grade 3; severe, Grade 4; life threatening
Severity of oral mucositis | For 21 days from the beginning of the chemotherapy
  Severity of oral mucositis was be evaluated by the World Health Organization Oral Toxicity Scale which record the extent and severity of oral mucositis every day.
  The World Health Organization Oral Toxicity Scale: range 0 to 4, Grade 0; none, Grade 1; mild, Grade 2; moderate, Grade 3; severe, Grade 4; life threatening
The duration of oral mucositis | From day 1 to day 21 of chemotherapy
  The duration of oral mucositis was be evaluated by the World Health Organization Oral Toxicity Scale which record the extent and severity of oral mucositis every day.
  The World Health Organization Oral Toxicity Scale: range 0 to 4, Grade 0; none, Grade 1; mild, Grade 2; moderate, Grade 3; severe, Grade 4; life threatening

SECONDARY OUTCOMES:
Time to onset of at least grade 2 oral mucositis | From day 1 to day 21 of chemotherapy
  Time to onset of at least grade 2 oral mucositis was be evaluated by the World Health Organization Scale which record the extent and severity of oral mucositis every day.
  The World Health Organization Oral Toxicity Scale: Grade 2; moderate, Grade 3; severe and Grade 4; life threatening
Time to onset of dry mouth | From day 1 to day 21 of chemotherapy
  Time to onset of dry mouth was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Incidence of dry mouth | For 21 days from the beginning of the chemotherapy
  Incidence of dry mouth was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Severity of dry mouth | For 21 days from the beginning of the chemotherapy
  Severity of dry mouth was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
The duration of dry mouth | For 21 days from the beginning of the chemotherapy
  The duration of dry mouth was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Time to onset of nausea | From day 1 to day 21 of chemotherapy
  Time to onset of nausea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Incidence of nausea | For 21 days from the beginning of the chemotherapy
  Incidence of nausea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Severity of nausea | For 21 days from the beginning of the chemotherapy
  Severity of nausea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
The duration of nausea | For 21 days from the beginning of the chemotherapy
  The duration of nausea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Time to onset of sensitivity/pain in the gums | From day 1 to day 21 of chemotherapy
  Time to onset of sensitivity/pain in the gums was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Incidence of sensitivity/pain in the gums | For 21 days from the beginning of the chemotherapy
  Incidence of sensitivity/pain in the gums was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Severity of sensitivity/pain in the gums | For 21 days from the beginning of the chemotherapy
  Severity of sensitivity/pain in the gums was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
The duration of sensitivity/pain in the gums | For 21 days from the beginning of the chemotherapy
  The duration of sensitivity/pain in the gums was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Time to onset of pain in the oral mucosa | For 21 days from the beginning of the chemotherapy
  Time to onset of pain in the oral mucosa was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Incidence of pain in the oral mucosa | For 21 days from the beginning of the chemotherapy
  Incidence of pain in the oral mucosa was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Severity of pain in the oral mucosa | For 21 days from the beginning of the chemotherapy
  Severity of pain in the oral mucosa was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
The duration of pain in the oral mucosa | For 21 days from the beginning of the chemotherapy
  The duration of pain in the oral mucosa was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Time to onset of dysphagia | For 21 days from the beginning of the chemotherapy
  Time to onset of dysphagia was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Incidence of dysphagia | For 21 days from the beginning of the chemotherapy
  Incidence of dysphagia was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Severity of dysphagia | For 21 days from the beginning of the chemotherapy
  Severity of dysphagia was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
The duration of dysphagia | For 21 days from the beginning of the chemotherapy
  The duration of dysphagia was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Time to onset of esophagitis | For 21 days from the beginning of the chemotherapy
  Time to onset of esophagitis was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Incidence of esophagitis | For 21 days from the beginning of the chemotherapy
  Incidence of esophagitis was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Severity of esophagitis | For 21 days from the beginning of the chemotherapy
  Severity of esophagitis was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
The duration of esophagitis | For 21 days from the beginning of the chemotherapy
  The duration of esophagitis was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Time to onset of diarrhea | For 21 days from the beginning of the chemotherapy
  Time to onset of diarrhea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Incidence of diarrhea | For 21 days from the beginning of the chemotherapy
  Incidence of diarrhea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Severity of diarrhea | For 21 days from the beginning of the chemotherapy
  Severity of diarrhea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
The duration of diarrhea | For 21 days from the beginning of the chemotherapy
  The duration of diarrhea was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 5, 1 was the mild, 5 was the death
Time to onset of weight loss | For 21 days from the beginning of the chemotherapy
  Time to onset of weight loss was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Incidence of weight loss | For 21 days from the beginning of the chemotherapy
  Incidence of weight loss was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
Severity of weight loss | For 21 days from the beginning of the chemotherapy
  Severity of weight loss was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe
The duration of weight loss | For 21 days from the beginning of the chemotherapy
  The duration of weight loss was be evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events Scale which to describe the severity of organ toxicity for patients receiving cancer therapy every day.
  The National Cancer Institute Common Terminology Criteria for Adverse Events Scale: Range 1 to 3, 1 was the mild, 3 was the severe

CONTACTS AND LOCATIONS:
Overall Officials: Seher ÇAKMAK Karadeniz Technical University, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)